CLINICAL TRIAL: NCT03152656
Title: A Registration Study for Familial Hypercholesterolemia in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201505031RIND
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2016-09

CONDITIONS: Familial Hypercholesterolemia
Keywords: Familial hypercholesterolemia; total cholesterol; low-density lipoprotein cholesterol; tendon xanthomas; premature atherosclerosis
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Familial hypercholesterolemia (FH) is an inherited disorder of lipoprotein metabolism, transmitted in an autosomal dominant manner and clinically characterized by elevated levels of total cholesterol (TC) and low-density lipoprotein (LDL) cholesterol, the presence of tendon xanthomas, and premature atherosclerosis.

The homozygous form of familial hypercholesterolemia (HoFH) with autosomal dominant transmission, in which case both alleles of either LDLR, APOB, or PCSK9 gene are defective, is a rare genetic disorder with prevalence estimated to be one per million population.

Large scale genetic screening for active FH cases finding has been performed in the Netherlands, Spain, Norway and Wales. However, the FH population and prevalence in Taiwan have never been formally studied. Patients are usually not under appropriate treatment owing to lack of standardized diagnostic tool and treatment strategy for FH. Moreover, with the emerging of new classes of LLTs, including microsomal triglyceride transfer protein (MTP) inhibitor, antisense oligonucleotide inhibitor, and PCSK9 inhibitors, even homozygous FH patients now have better chance to be treated to reach recommended treatment goals. Therefore, A National FH registry is needed to collect contemporary data on diagnosis, treatment and outcomes with long- term goals of improving diagnosis, management, and reduction of unnecessary cardiovascular events in FH population in Taiwan.

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is an inherited disorder of lipoprotein metabolism, transmitted in an autosomal dominant manner and clinically characterized by elevated levels of total cholesterol (TC) and low-density lipoprotein (LDL) cholesterol, the presence of tendon xanthomas, and premature atherosclerosis.The genetic basis of FH is a large array of point mutations and large gene rearrangements in the LDL receptor (LDLR) gene, resulting in defective functional receptors for LDL on the cell surface, which are unable to clear plasma LDL and result in increased plasma LDL levels. Similarly, point mutations in the gene coding for apolipoprotein B (APOB) also reduce LDL clearance, resulting in the disorder familial defective apolipoprotein B, which is clinically indistinguishable from FH. In 2003, a third FH locus located on chromosome 1, encoding proprotein convertase subtilisin/kexin 9 (PCSK9) was identified. The phenotypes caused by mutations in LDLR, APOB, or PCSK9 are clinically indistinguishable and all characterized by elevated levels of plasma LDL cholesterol and premature coronary artery disease.

The homozygous form of familial hypercholesterolemia (HoFH) with autosomal dominant transmission, in which case both alleles of either LDLR, APOB, or PCSK9 gene are defective, is a rare genetic disorder with prevalence estimated to be one per million population. Patients with HoFH have an extremely rapid accumulation of atherosclerosis with most experiencing xanthomas and severe vascular disease by adolescence or early adulthood despite interventions, including LDL apheresis, which led to the recent Food and Drug Administration approval of 2 novel therapies, lomitapide and mipomersen, specifically for HoFH. Heterozygous familial hypercholesterolemia (HeFH), in which only one allele of LDLR, APOB or PCSK9 gene is defective, has a prevalence of approximately one in 500 individuals, making it one of the most common inherited disorders. Reduction of elevated cholesterol levels in FH individuals can result in a significant reduction of cardiovascular mortality and morbidity, as a large number of landmark clinical trials with cholesterol synthesis inhibitors have clearly demonstrated. However, less than 10% of patients with HeFH are diagnosed and less than 25% are treated with LDL-lowering medications.

Large scale genetic screening for active FH cases finding has been performed in the Netherlands, Spain, Norway and Wales. However, the FH population and prevalence in Taiwan have never been formally studied. Patients are usually not under appropriate treatment owing to lack of standardized diagnostic tool and treatment strategy for FH. Moreover, with the emerging of new classes of LLTs, including microsomal triglyceride transfer protein (MTP) inhibitor, antisense oligonucleotide inhibitor, and PCSK9 inhibitors, even homozygous FH patients now have better chance to be treated to reach recommended treatment goals. Therefore, A National FH registry is needed to collect contemporary data on diagnosis, treatment and outcomes with long- term goals of improving diagnosis, management, and reduction of unnecessary cardiovascular events in FH population in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Taiwan FH Diagnostic Criteria was revised from Dutch Lipid Clinic Network (DLCN) Criteria with consensus of experts in cardiology, genetic, and metabolism specialty, and published by Taiwan Society of Lipids & Atherosclerosis in 2014.

Exclusion Criteria:

* The main exclusion criteria will be secondary causes of hyperlipidemia other than FH (i.e. untreated hypothyroidism, nephrotic syndrome), hemodynamically significant valvular or congenital heart disease, life-threatening malignancy, treatment with immunosuppressive agents, or any condition or situation which, in the opinion of the investigator, might be not suitable for this registration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potentially eligible patients will be invited for a screening visit. Written informed consent will be obtained from all patients, and the study will be approved by the institutional review board.
  1000 Subjects (estimated) with diagnosis of definite or probable FH, including both heterozygous and homozygous FH, using Taiwan FH Diagnostic Criteria will be recruited for enrollment and clinically followed for at least three years. Taiwan FH Diagnostic Criteria was revised from Dutch Lipid Clinic Network (DLCN) Criteria with consensus of experts in cardiology, genetic, and metabolism specialty, and published by Taiwan Society of Lipids & Atherosclerosis in 2014.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Composite cardiovascular outcome | 3 years
  The composite cardiovascular (CV) outcome will be any CV events (coronary, cerebral, or peripheral vascular diseases)

SECONDARY OUTCOMES:
With at least 1 cardiovascular risk factor. | 3 years
  no evidence of atherosclerotic vascular diseases,with at least 1 cardiovascular risk factor.

CONTACTS AND LOCATIONS:
Overall Officials: Chau C Wu, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes